CLINICAL TRIAL: NCT05022225
Title: Psychosocial Reasons for Transfer to In Center Hemodialysis in Home Dialysis Patients- A Focus Group Study
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: SIH128_Transfer to ICHD
Record Dates: First submitted 2021-08-13; First posted 2021-08-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: ESRD
Keywords: home dialysis; Peritoneal dialysis; home hemodialysis; patient perspective
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None. This is a qualitative interview study. — There is no intervention in this study. This is a qualitative research study where participants will take part in focus group discussions.

SUMMARY:
Patients who start home dialysis take on an added responsibility and that can be challenging. The investigators are interested in studying the patient and care partner perspective on the challenges that the participants faced on home dialysis and what interventions could help support them better by holding focus group discussions.

DETAILED DESCRIPTION:
Home dialysis has many advantages compared to in-center hemodialysis (ICHD) including better quality of life and lower healthcare costs. Transfer from home dialysis to ICHD is disruptive to the patients' lives and in some cases may be preventible. Patients do not infrequently transfer to ICHD due to psychosocial reasons, which may be multi-factorial and hard to capture.

The aim of this study is to explore patients' and care partners' perspectives and experiences of the psychosocial factors that make home dialysis challenging and that ultimately contribute to transfer to ICHD during focus group discussions. The investigators will ask them to describe issues that may compound patient and care partner burnout; for those who have already transferred to hemodialysis, the investigators will specifically ask what factors contributed to their transfer off of home dialysis. the investigators will also ask for feedback on what interventions may have helped to prevent the transfer and/or burnout.

* Understanding patient's perspectives and experiences will help the investigators improve patient experience and identify the gaps in health care delivery.
* Help plan interventions and scale-out a solution to identify patients experiencing challenges that put them at risk of transfer to ICHD.
* Lay the groundwork to develop surveys that can be used in the future.
* To enable a truly patient-centered care model, understanding the issues in more detail is critical.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently on home dialysis (maintenance peritoneal dialysis or home hemodialysis), preferably identified as high risk of transfer to in center HD at Satellite healthcare by the clinical team, OR their care partner
* Patients who transferred from home dialysis to ICHD in the last 12 (preferably 6) months, preferably those who had transferred mostly because of psychosocial reasons such as nonconducive living conditions, patient preference, the burden of treatment, loss of care partner, etc, OR their care partner.
* Age >=20 years

Exclusion Criteria:

* Lack of decision-making capacity
* Non English-speaking

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients at Satellite health care who transferred to ICHD from home dialysis in the last year and home dialysis patients who are identified as high risk for transfer to ICHD by the clinical team.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Patients and care partner experience on home dialysis | At the time of focus group discussion
  During the focus group discussion, the participants will be asked to account their experience on home dialysis and the challenges that they faced while on the modality. Since it is a qualitative study the responses will be grouped to identify any common themes.

SECONDARY OUTCOMES:
patient and care partner perspective on possible interventions | At the time of the focus group discussion
  During the focus group discussion the participants will be asked if there were any interventions that were offered or if there are any interventions that would have helped support them better on home dialysis. Since it is a qualitative study the responses will be grouped to identify any common themes.
comparison between groups | At the time of focus group
  Different themes between the participant responses will be compared after a thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Wael F Hussein, MBBS, Principal Investigator — Satelite Health care
Locations (1):
- Satellite Healthcare Inc, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No
No individual person data will be available to anyone other than Satellite Healthcare Research employees.